CLINICAL TRIAL: NCT01781910
Title: The Effects of Branched Chain Amino Acid and Nutrient Supplementation on Exercise-Induced Delayed Onset Muscle Soreness in College Females
Brief Title: Branched Chain Amino Acid Plus Glucose Supplement Reduces Exercise-Induced Delayed Onset Muscle Soreness in College Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Stephen J. Pintauro, Associate Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHRMS M12-101
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Exercise-induced Delayed Onset Muscle Soreness
Keywords: branched chain amino acids, exercise, delayed onset muscle soreness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Branch Chain Amino Acid supplement (Experimental): A drink supplement containing 1.22 grams of branched chain amino acids, plus glucose.
  Interventions: Dietary Supplement: Branched Chain Amino Acid drink supplement
- Placebo supplement (Placebo Comparator): The placebo was formulated to match both the taste and color of the test supplement. Crystal Light Lemonade powder (Kraft Foods, Northfield, IL, USA) was mixed with 5.6g of powdered dextrose (Now Foods, Bloomingdale, IL, USA) to match the amount of dextrose present in the BCAA supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Branched Chain Amino Acid drink supplement
  Arms: Branch Chain Amino Acid supplement
Dietary Supplement: Placebo
  Arms: Placebo supplement

SUMMARY:
The purpose of this study is to determine if a dietary supplement containing branched chain amino acids will reduce the muscle soreness that sometimes occurs in the days following exercise.

DETAILED DESCRIPTION:
Supplementation with branched chain amino acids (BCAAs) has been used to stimulate muscle protein synthesis following exercise. The purpose of this study was to determine if supplementation with BCAAs in combination with glucose would reduce exercise-induced delayed onset muscle soreness (DOMS). Using a double-blind crossover design, 20 subjects (11 females, 9 males) were randomly assigned to either BCAA (n=10) or placebo (n=10) groups. Subjects performed a squatting exercise to elicit DOMS and rated their muscle soreness every 24 hours for four days following exercise while continuing to consume the BCAA or placebo. Following a three-week recovery period, subjects returned and received the alternate BCAA or placebo treatment, repeating the same exercise and DOMS rating protocol for the next four days. BCAA supplementation in female subjects resulted in a significant decrease in DOMS versus placebo at 24 hours following exercise (p = 0.018). No significant effect of BCAA supplementation versus placebo was noted in male subjects, nor when male and female results were analyzed together. This gender difference may be related to dose per body weight differences between male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men (n=9) and women (n=11) aged 18-25 who engaged in no more than one hour of light to moderate intensity physical activity per week were recruited from the Greater Burlington, Vermont area.

Exclusion Criteria:

* individuals who engaged in more than one hour per week of light to moderate physical activity
* had been involved in strict athletic competition or weight training in the past six months
* were pregnant or nursing, had a known muscular disease, diabetes mellitus, cardiovascular disease, respiratory disease, and/or were currently taking a protein-based dietary supplement

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Delayed Onset Muscle Soreness Rating Scale | Every 24 hours for four days following exercise

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Pintauro, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States